#### Makerere University Walter Reed Project

#### INFORMED CONSENT FOR OPTIONAL LYMPH NODE BIOPSY

**Title of Protocol:** A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to

Evaluate the Safety, Tolerability, and Immunogenicity of an

Ad26.Mos4.HIV and CH505 TF chTrimer (Env) Combination to Mimic

Acute HIV Viral Replication Kinetics in Healthy Adults

**Sponsor:** The Surgeon General, Department of the Army

**Principal** 

**Investigator:** Grace Mirembe, MBChB, MMed

#### Introduction

The purpose of this consent form is for study participants to indicate their willingness to participate in the optional lymph node biopsy procedure for this study and if you will allow us to photograph the incision site. Before you decide whether to take part in this procedure and whether you will allow photos to be taken, we would like to explain the purpose, how it may help you or others, any benefits and risks associated with the procedure, and our expectations of you.

Please read this form carefully. If you have any questions or concerns about the optional lymph node biopsy procedure, about the photographs of the incision site, or about this form, please ask us. You can take as much time as you need to review this form and discuss your participation with your family, friends, and community as you feel comfortable and as appropriate in order to decide whether you would like to participate in the optional procedure and have pictures taken. You will be given as much time as you need to make this decision. Taking part in the optional lymph node biopsy procedure as well as the decision to allow photographs is up to you and you will still be allowed to participate in this study if you choose not to participate in the optional lymph node biopsy procedure and/or refuse to allow pictures to be taken. Whether or not you decide to take part in the optional lymph node biopsy procedure or allow photos, you must mark your choices at the end of the form as well as sign this form. We will give you a signed copy of this form to keep.

The optional lymph node biopsy procedure is for research and not for treatment. The photographs are also optional and are not required for participation in the lymph node biopsy. It is possible that some people who consent to the optional lymph node biopsy procedure may not be selected to have it performed. This will in no way affect your participation in the main study. There will be no negative consequences to you if you decide not to take part in the optional lymph node biopsy procedure or if you refuse to allow photos to be taken.

# What do I need to know about the optional lymph node biopsy procedure? We would like you to know the following:

1. The optional lymph node biopsy procedure may be done on the same day as your Visit 7 (Study Day 71) for the main study or on a different day (within 7 days after the main study visit). Researchers will try to accommodate your preference as much as possible.

- 2. The optional lymph node biopsy procedure will be completed by trained medical personnel at Case Medical Center (also known as Case Hospital). Study staff will make an appointment for you to have the biopsy completed if you choose to undergo the procedure.
- 3. For female participants, you will not be eligible to undergo the optional lymph node biopsy procedure if you are pregnant as it may cause unforeseeable risk to you and/or your fetus. You will be tested for pregnancy before the procedure to ensure that you are not pregnant.
- 4. For your safety, you will not be able to undergo the optional lymph node biopsy procedure if the results from the pre-biopsy safety tests indicate that you are at an increased risk for bleeding, you have a bleeding or blood clotting disorder, you cannot safely stop taking certain medications prior to the procedure, you have previously had 4 or more lymph nodes removed at any time in your life, or you will not receive any further study injections.
- 5. If you undergo the optional lymph node biopsy procedure and there is evidence of an abnormal finding, you will be referred for diagnosis and care.

### What is a biopsy?

A biopsy is a procedure where body tissue is removed to test for disease. In this study, we will store the biopsy samples to study your body's response to the vaccine.

### What is a lymph node?

Lymph nodes are small natural nodules that are a part of your immune system and can be found behind the ears, in the neck, in the armpit, and in the groin. Lymph nodes are responsible for producing some white blood (immune) cells called lymphocytes as well as filtering the fluid that carries them around in the body. They usually swell when you have an infection nearby (e.g., a wound on the leg can cause the lymph node in your groin to swell).

## Why is a lymph node biopsy done?

The body's defenses against HIV infection are not well understood. Two of the main types of cells that are important in the body's immune system, the T cells and the B cells, are found in large numbers within your lymph nodes. In the future, to try to develop better treatments for and vaccinations against HIV, it is important for us first to understand the interactions between these cells, their roles in immunity and how these are affected by HIV infection and HIV treatment.

# How is a lymph node biopsy done?

A surgeon will perform the lymph node biopsy under local anesthetic. This means you will be awake, but the biopsy area will be numb. The surgeon will biopsy a lymph node in the groin area because this is the safest location with the smallest risk of problems. The surgeon will clean your groin with an antiseptic solution and then make a small cut in the groin (about 1 to 2 centimeters long). The surgeon will remove a lymph node, which is about the size of a peanut, through the incision. The surgeon will then close the incision with absorbable stitches and bandage the wound. The whole process will take about 30 to 40 minutes. You will remain under observation for up to 4 hours after the procedure. You will also be asked not to do any strenuous activities for the next 24 hours. The study staff will call to follow up with you about 3 to 4 days after procedure to see if there are any problems.

With your permission, we would like to take pictures of the wound right after the procedure, 2 weeks after the procedure, and 3 months after the procedure to follow the wound healing. The pictures taken at 2 weeks and 3 months post-procedure will be completed at your scheduled study visit. Researchers may use these pictures as educational material for other subjects who are interested in undergoing the same procedure. You must indicate your decision at the end of this form. You are free to decline the photography and still undergo the procedure. Refusal to have these photographs taken will not have any effect on your study participation. We will make an effort to avoid photographing your face, any tattoos, or any birthmarks that could be used to identify you in the photo. Your name and other identifying information will not be associated with the photograph. All photographs will be the property of the site. Photographs will relate only to this study.

### What are the benefits of the optional lymph node biopsy procedure?

You may benefit from the additional medical screening and subsequent treatment referrals in the event that there are any abnormal findings. Other than the screening and referrals for treatment, you will not gain any direct benefit from participating in the optional lymph node biopsy procedure, however the results of this study will provide important information on the design of vaccines to prevent HIV, including possible improvements to future vaccines and timeline for development. Data collected from this study will be used to further develop a vaccine to prevent HIV. If this study vaccine or related vaccines can prevent HIV infection, this could benefit the general population.

### What are the risks of the optional lymph node biopsy?

You may experience pain in the biopsy area once the local anesthetic has worn off. If you have pain, the study team will provide additional medications to control the pain. There is the possibility of some bleeding following the procedure. Doctors will perform blood tests before the biopsy and ask about any medications you are taking or conditions you have that may make you more likely to bleed. You should not take certain drugs such as aspirin and anti-inflammatory drugs (the investigator will explain this to you) for 7 days before the procedure. For your safety, you will not be able to undergo the procedure if the results from the pre-biopsy safety tests indicate that you are at an increased risk for bleeding, you have a bleeding or blood clotting disorder, or you cannot safely stop taking medications for 7 days before the procedure.

The procedure will be performed using sterile equipment, but there is still a small risk of infection. If the doctor who reviews the wound feels that it is infected, the doctor will provide you with antibiotics to treat the infection. It is also possible that you may develop fluid filled swelling in the area of the biopsy, which may require drainage or further management, or nerve damage which could result in temporary or permanent loss of feeling in the biopsy area. If you have any concerns that your wound might be infected, that there may be some fluid filled swelling, or that you have lost some feeling in the biopsy area, you should contact the study team for further management or a referral for care and treatment. You may also notice bruising around the area of the biopsy and there is the possibility of developing a scar as the wound heals. These risks are minimized by the small size of the cut from which a lymph node will be taken out.

It is possible, although unlikely, that the surgeon will be unable to find a lymph node or for some reason unable to remove it during the procedure. In that case, the procedure will be stopped without removing a lymph node.

There is a small risk of chronic swelling of the leg on the side that the lymph node is taken from. For this reason, it is recommended that one participant have no more than 4 inguinal lymph node biopsies, or 2 biopsies per side, done in their entire life, which would include this study, any other studies that collect a lymph node, and any medical procedures performed elsewhere for non-research purposes.

After the procedure, you may feel dizzy, sleepy, confused or nauseated from the anesthetic and pain medicines; therefore, you should have someone come with you to accompany you home. There is a very small risk for a more severe allergic reaction to the anesthetic. You should not drive a vehicle after the procedure.

### How often is a lymph node biopsy done?

The lymph node biopsy will happen 1 time during the study: at or within 7 days after Visit 7 (Study Day 71).

### How long will my lymph node biopsy samples be stored?

If you have given your permission for the storage of your biological samples in the "Future Use of Stored Specimens" informed consent form, your lymph node tissue will be stored indefinitely. The samples will not be labelled with any personal information, such as your name. Instead, they will have your study code. The link between your personal information and your study code will be kept secure with access limited to only those who need the information to conduct the study. If you have not given your permission for the storage and future use of your samples, they will be used as described for this study and then destroyed at the end of the study.

# Do I have other options?

You may decide not to take part in the optional lymph node biopsy procedure and still take part in the main study.

## **Early termination**

The optional lymph node biopsy procedure may be stopped early or not done at all if the investigators feel that it is causing you harm or if the sponsor decides to stop the study.

# Confidentiality

The researchers will maintain the confidentiality of your personal information and will not release this information without your express permission or unless required by the law. In order to ensure that the study is being run appropriately and ethically, other bodies (for example the sponsoring organization, Institutional Review Board or drug licensing authorities) may also exercise the right to access, verify or audit study information, including the personal information of study participants. By joining this study, you also give permission for information, which may include your medical records, to be accessed.

### What are the costs to you?

You will not have to pay for any of the study procedures. The study team will support costs related to your participation.

### Will I get any payment for transportation and loss of time?

If you consent to participate in the optional lymph node biopsy, you will receive Ug shs 70,000 for a pre-lymph node biopsy safety blood draw visit and Ug shs 200,000 as compensation for your time, transportation, and inconvenience associated with the procedure. You will receive this compensation even if the safety blood draw is completed during a scheduled visit or the surgeon is unable to find or remove a lymph node.

The compensation amounts listed above are in addition to the compensation that you will receive for the main study visits. You will receive compensation for the main study even if you don't take part in the optional lymph node biopsy procedure.

### What will happen if I am injured?

If you get sick or injured as a result of the study procedures, you will receive appropriate medical treatment and care until cure or stabilization as provided for by a limited fund (set aside for this study) and a clinical trials medical insurance policy for research-related injuries. While we anticipate the combination of the set-aside fund and the insurance policy is more than enough to pay for the costs associated with any study related injuries, there is a limit to the amount of coverage available. The study sponsor, MUWRP, and the U.S. DoD will not provide long-term medical care for stabilized research-related injuries.

The study team is responsible for the cost without using any personal health care package which belongs to you. MUWRP will pay costs up to the limit from set aside finds or through the insurance. However, you will not receive any other compensation. You should discuss this thoroughly with the Principal Investigator or site clinicians before making a decision to participate in this optional procedure.

#### For more information:

If you have questions about the optional lymph node biopsy procedure, a problem that you think may be related to the optional lymph node biopsy procedure, or if you want to withdraw your consent, you can contact Dr. Grace Mirembe by telephone at 0312-330400, 0800-200058, or 0772-577768; or you can contact the study coordinator, Dr. Job Kasule by telephone at 0312-330400, 0800-200058, or 0701-772291.

If you have questions about your rights as a research participant, problems or concerns about how you are being treated in this study, or feel that you have not received the appropriate care and treatment for a sickness or injury that occurred as a direct result of taking part in this study, you may contact Dr. Joseph Kagaayi at the Research and Ethics Committee, Makerere University School of Public Health, Mulago Hospital Complex by telephone at 0773-785333 or you may contact The Executive Secretary at the Uganda National Council for Science and Technology by telephone at 0414-705500.

#### INFORMED CONSENT FOR OPTIONAL LYMPH NODE BIOPSY

"A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of an Ad26.Mos4.HIV and CH505 TF chTrimer (Env) Combination to Mimic Acute HIV Viral Replication Kinetics in Healthy Adults"

### **Participant Statement:**

**Lymph Node Biopsy** 

The principal investigator, Dr. Grace Mirembe or their representative has explained in detail the purpose of the optional lymph node biopsy, the purpose of the incision site photographs, the procedures involved, and the risks and benefits of the procedure. I have been informed that by signing this form, I am not giving up any legal rights. I have been given a chance to ask questions about the lymph node biopsy procedure as well as the incision site photographs, and all of my questions were answered to my satisfaction. If I have other questions about this study, I can contact Dr. Grace Mirembe, by telephone at 0312-330400, 0800-200058, or 0772-577768; or I can contact the study coordinator, Dr. Job Kasule by telephone at 0312-330400, 0800-200058, or 0701-772291.

I am indicating my decision of whether to participate in the option lymph node biopsy procedure and whether to allow photographs to be taken of the incision site by marking the applicable boxes below, writing my initials next to the marked boxes, and printing and signing my name in the spaces provided below. I will do my best to follow the recommendations of the study team, and I will report all problems occurring from this study to the study team. It has been explained to me that even if I agree to the procedure now, I have a right to end my participation in the optional lymph node biopsy procedure at any time and without losing any rights to which I am entitled. The medical care that I could receive as a result of any sickness or injury that may result from being a part of this study have been explained to me and I have been offered a signed copy of this consent form.

# I agree to undergoing the optional lymph node biopsy procedure. The procedure initials has been explained to me and all of my questions have been answered to my satisfaction. The risks of the procedure have also been explained to me. I understand that in addition to the risks described to me about this procedure, there are risks that may occur with any medical procedure. I do not agree to undergoing the optional lymph node biopsy procedure. initials **Incision Site Photographs** I allow photographs to be taken of the lymph node biopsy incision site. I have initials been informed that the investigators will try not to include my face, tattoos, or birthmarks that could be used to identify me. I have been given the opportunity to ask questions and all of my questions have been answered to my satisfaction. I do not agree to having photographs taken of the lymph node biopsy incision site. initials

| SIGNATURE OF PARTICIPANT | DATE |
|--------------------------------------------|------|
| PRINT NAME OF PARTICIPANT | |
| SIGNATURE OF PERSON ADMINISTERING CONSENT | DATE |
| PRINT NAME OF PERSON ADMINISTERING CONSENT | |